CLINICAL TRIAL: NCT05262855
Title: A Phase 2, Multicenter, Single Arm, Open Label Non-Randomized Study of [68Ga]FAPI-46 PET in Patients With Resectable or Borderline Resectable Pancreatic Ductal Carcinoma
Brief Title: Study of [68Ga]FAPI-46 PET in Patients With Pancreatic Ductal Carcinoma
Acronym: FAPI-46 PDAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SOFIE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GaFAPI-2022P2
Record Dates: First submitted 2022-02-10; First posted 2022-03-02 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: PDAC - Pancreatic Ductal Adenocarcinoma; FAP
Keywords: Fibroblast Activation Protein Inhibitor (FAPI); PDAC
MeSH Terms: interventions — FAPI-46

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI-46 PET/CT (Experimental): Patients receive [68Ga]FAPI-46 intravenously followed by PET/CT 15-25 minutes later
  Interventions: Drug: [68Ga]FAPI-46

INTERVENTIONS:
Drug: [68Ga]FAPI-46 — [68Ga]-FAPI-46 is a radioactive diagnostic agent indicated for use with Positron Emission Tomography (PET) imaging for the detection of Fibroblast Activation Protein (FAP) positive cancer cells and cancer-associated fibroblasts (CAF) in patients with pancreatic ductal adenocarcinoma (PDAC).

SUMMARY:
This is a prospective, multi-center, single arm, open label, non-randomized study to evaluate the ability of [68Ga]FAPI-46 to detect FAP expressing cells in patients with resectable or borderline resectable PDAC. The [68Ga]FAPI-46 PET scans will be acquired after initial staging using institutional standard methods. If the participant is prescribed neoadjuvant therapy, a second [68Ga]FAPI-46 PET scan will be performed within 21 days prior to planned surgical resection. This will be followed by histopathology and IHC analyses and comparison to resected PDAC tumor specimens.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed pancreatic ductal adenocarcinoma
2. Treatment-naïve
3. Staged as resectable or borderline-resectable
4. Planned to undergo surgical resection or to receive neoadjuvant therapy (i.e., chemotherapy, radiation therapy, or combination) and subsequent possible surgical resection
5. Anatomic imaging (e.g., CT, MRI) obtained within ≤ 28 days of consent
6. Age ≥ 18 years
7. Completed informed consent as determined per the IRB of record

Exclusion Criteria:

1. Pregnant as determined by a pregnancy test as per institutional guidelines for individuals of child-bearing potential
2. Declining to use effective contraceptive methods during the study (for individuals of child-producing potential)
3. Need for emergent surgery that would be delayed by participation
4. Bacterial, viral, or fungal infections requiring systemic therapy
5. Serious co-morbidities and serious nonmalignant disease (e.g., hydronephrosis, kidney failure, liver failure, systemic or local inflammatory or autoimmune diseases or other conditions) that in the opinion of the investigator, physician of record and/or Sofie could compromise patient safety and/or protocol objectives.
6. Known diagnosis of autoimmune disorders
7. Patients receiving any other investigational agent within the past 28 days
8. Breastfeeding. Note: nursing parents are allowed if the potential participant commits to pumping breast milk and discarding it from injection to ≥ 24 hours from the time of the [68Ga]FAPI-46 injection.
9. Known hypersensitivity to any excipients used in [68Ga]FAPI-46:

trace amounts of sodium acetate sodium ascorbate and/or hydrochloric acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Performance [sensitivity, specificity, accuracy] of [68Ga]FAPI-46 PET imaging to detect FAP-expressing cells, using histopathology as truth standard. | Through study completion, 2 years

SECONDARY OUTCOMES:
Positive and negative predictive values, as well as accuracy of [68Ga]FAPI-46 PET images, to detect FAP-expressing cells using histopathology as truth standard. | Through study completion, 2 years
Histopathology with FAP staining on FAP IHC assay. | Through study completion, 2 years
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to 24 hours post injection with [68Ga]FAPI-46
[68Ga]FAPI-46 accumulation observed in local and metastatic disease compared to radiological (i.e. CT, MR) and/or 18F-FDG PET. | Through study completion, 2 years
[68Ga]FAPI-46 accumulation observed by (PET)/ (CT) pre and post in patients undergoing Neoadjuvant treatment. | Through study completion for patient undergoing Neoadjuvant treatment, 2 years

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of California Los Angeles (UCLA) Health, Los Angeles, California
  - BAMF Health, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Karbhari A, Mosessian S, Trivedi KH, Valla F Jr, Jacobson M, Truty MJ, Patnam NG, Simeone DM, Zan E, Brennan T, Chen H, Kuo PH, Herrmann K, Goenka AH. Gallium-68-labeled fibroblast activation protein inhibitor-46 PET in patients with resectable or borderline resectable pancreatic ductal adenocarcinoma: A phase 2, multicenter, single arm, open label non-randomized study protocol. PLoS One. 2023 Nov 27;18(11):e0294564. doi: 10.1371/journal.pone.0294564. eCollection 2023. PMID 38011131